## Quantitative Electroencephalogram (QEEG) Predictors of Response to Psychotherapy Versus Antidepressant Treatment in Depression

Identifiers: NCT00824044

Unique Protocol ID: 2008-P-000838

Date prepared: 12/7/2017

## Summary:

A-priori expectation from prior **medication** work is a decrease in theta activity from baseline at week 1 in responders, and an increase in non-responders. Prior work showed an increase in theta activity in **placebo** responders (and little change in non-responders). (See attached manuscript that describes changes in theta Cordance over time in both placebo and medication groups. See Fig 4 on page 128.) Also, ATR is expected to be higher in medication responders than non-responders after 1 week on antidepressant.

## Methods:

ATR and Power metrics were calculated from available EEGs at baseline and subsequent visits. Change in Power between baseline and subsequent visits were derived. The data were analyzed for 3 groups: Pooled, Drug-only, Drug+CBT.

In a completer analysis (not an intent to treat), independent sample t tests were used to assess the relationship between responders (greater than or equal to 50 % reduction in the primary outcome (HAMD-17 score)) and change in QEEG metrics across time.